CLINICAL TRIAL: NCT02888080
Title: A Multiple-dose, Subject and Investigator Blinded, Placebo-controlled, Parallel Design Study to Assess the Efficacy, Safety and Tolerability of ACZ885(Canakinumab) in Patients With Pulmonary Sarcoidosis
Brief Title: Study of Efficacy, Safety and Tolerability of ACZ885 (Canakinumab) in Patients With Pulmonary Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CACZ885X2205
Record Dates: First submitted 2016-08-16; First posted 2016-09-02 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Sarcoidosis
Keywords: pulmonary sarcoidosis; sarcoidosis; canakinumab; autoimmune diseases; granulomas; inflammation; lung function testing; immunosuppressive agents; interleukin; interleukin-1Beta; [F-18]FDG-PET/CT; respiratory; pulmonary; steroids; corticosteroids; lung diseases
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis; Autoimmune Diseases; Granuloma; Inflammation; Lung Diseases | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACZ885 (Experimental): ACZ885 (300 mg/2 mL) will be administered subcutaneously to assigned study subjects once monthly for 6 months.
  Interventions: Drug: ACZ885
- Placebo (Placebo Comparator): Placebo (0 mg/2 mL) will be administered subcutaneously to assigned study subjects once monthly for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACZ885 — ACZ885 will be administered subcutaneously to assigned study subjects once monthly for 6 months.
  Other Names: Canakinumab
  Arms: ACZ885
Drug: Placebo — Placebo will be administered subcutaneously to assigned study subjects once monthly for 6 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if ACZ885 will improve lung function in association with reduction of tissue inflammation in patients with chronic sarcoidosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects ages 18 to 80 years of age (both inclusive)
* Pulmonary sarcoidosis disease duration of ≥1 year
* Clinically active disease demonstrated either by a biopsy (any organ) or by bronchoalevolar lavage (lymphocytosis >15%, CD4+/CD8+ ration>3.5, CD103+/CD4+/CD4+ ratio <0.2). Patients must also have all of the following criteria:

  1. MMRC dyspnea scale ≥1
  2. Threshold FVC 50 - 90% of predicted
  3. Evidence of parenchymal lung involvement by HRCT at screening or by historical radiological evidence (e.g. CT, MRI or x-ray)

Key Exclusion Criteria:

* Treated pulmonary hypertension
* Previous exposure to concomitant treatment according to the following criteria:

  1. Prednisone >15 mg/day or changes in prednisone dose in the 8 weeks prior to screening
  2. More than one immune-modulator (i.e., methotrexate, azathioprine, leflunomide, hydroxychloroquine) or changes in their dosing levels within 12 weeks of randomization.
  3. Mycophenolate use within 12 weeks of randomization
* Prior treatment with any biologic drug targeting the immune system within 180 days of randomization or history of any previous use of rituximab
* History of bleeding disorder
* Forced vital capacity (FVC) <50% of predicted
* Extra-pulmonary sarcoidosis as primary treatment indication (e.g., involving brain, heart, eye and renal disease with significant hypercalcemia)
* Any conditions or significant medical problems which in the opinion of the investigator immune-compromise the patient and/or places the patient at unacceptable risk for immunomodulatory therapy, such as:

  1. Absolute neutrophil count (ANC) <LLN (1,500/μl)
  2. Thrombocytopenia CTCAE v4.03 Grade 1: Platelets <LLN (75.0 x 10exp9/L)
  3. Any active or recurrent bacterial, fungal (with exception of onychomycosis) or viral infection
  4. Presence of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C infections based on screening lab results
  5. Presence of active or latent tuberculosis (Tb). If historical Tb result is available, Tb status needs to be confirmed pre-randomization as determined by screening laboratory measurements.
  6. Clinical evidence or history of multiple sclerosis or other demyelinating diseases, or Felty's syndrome
* Live vaccinations within 3 months prior to the start of the trial
* Current severe progressive or uncontrolled disease which in the judgment of the clinical investigator renders the patient unsuitable for the trial
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using methods of contraception defined in the protocol for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Cleveland, Ohio
- Germany (3):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hanover
- Netherlands (2):
  - Novartis Investigative Site, Nieuwegein
  - Novartis Investigative Site, Rotterdam

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=499

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety Analysis set : 20 patients ACZ885 and 20 patients Placebo
  PK Analysis set : 20 patients ACZ885
  PD Analysis set : 20 patients CAZ885 and 20 patients placebo
Groups:
- ACZ885: ACZ885 (300 mg s.c. once monthly for 6 months)
- Placebo: Placebo (s.c. once monthly for 6 months)
Period: Overall Study
Arm/Group | ACZ885 | Placebo
Started | 20 | 20
Completed | 18 | 15
Not Completed | 2 | 5
Not completed — Subject / Guardian decision | 1 | 3
Not completed — New Therapy for study indication | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACZ885 | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (8.45) | 48.1 (9.94) | 50.0 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 12 | 16 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Black or African American | 2 | 1 | 3
    White | 18 | 16 | 34
    Asian | 0 | 2 | 2
    Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change Between Baseline and Week 24 in Pulmonary Function as Measured by Spirometry
Description: To compare the effect of ACZ885 versus placebo in the change between baseline and week 24 in pulmonary function as measured by spirometry (Predicted Forced Vital Capacity).
Time Frame: Baseline, Week 24
Population: Pharmacodynamic Analysis Set, with measure
Measure: Mean (Standard Deviation); unit: Percent Predicted Forced Vital Capacity
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
Percent Predicted Forced Vital Capacity | -1.90 (3.91) | 0.52 (3.37)

2. Secondary Outcome: Change Between Baseline and Week 12 in Pulmonary Tissue Inflammation (Lung Parenchyma) as Measured by SUVmax[F-18]FDG-PET/CT
Description: To determine the effect of ACZ885 on the change of pulmonary tissue inflammation as measured by SUVmax[F-18]FDG-PET/CT from baseline after 12 weeks of treatment compared to placebo.
Time Frame: Baseline, Week 12
Population: Pharmacodynamic Analysis Set, with measure
Measure: Mean (Standard Deviation); unit: percentage (Mean % Change In SUVmax)
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
percentage (Mean % Change In SUVmax) | -4.48 (37.45) | 4.07 (26.61)

3. Secondary Outcome: Change Between Baseline and Week 12 in Nodular Uptake Regions as Measured by SUVmax[F-18]FDG-PET/CT
Description: To determine the effect of ACZ885 on decreasing the maximum standardized uptake value (SUVmax) [F-18]FDG-PET in nodules (nodular uptake regions) after 12 weeks of treatment, compared to placebo.
Time Frame: Baseline, Week 12
Population: Pharmacodynamic Analysis Set, with measure
Measure: Mean (Standard Deviation); unit: percentage (Mean % Change In SUVmax)
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
percentage (Mean % Change In SUVmax) | -7.70 (35.77) | 1.03 (41.10)

4. Secondary Outcome: Change Between Baseline and Week 12 in in the Extrathoracic Region as Measured by SUVmax[F-18]FDG-PET/CT
Description: To determine the effect of ACZ885 on decreasing the maximum standardized uptake value (SUVmax) [F-18]FDG-PET in in the extrathoracic Region after 12 weeks of treatment, compared to placebo.
Time Frame: Baseline, Week 12
Population: Pharmacodynamic Analysis Set, with measure
Measure: Mean (Standard Deviation); unit: percentage (Mean % Change In SUVmax)
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
percentage (Mean % Change In SUVmax) | -21.4 (13.15) | 1.76 (39.60)

5. Secondary Outcome: Change From Baseline in Other Parameters of Pulmonary Function Testing (FEV 1, 3, 6 Seconds and Predicted)
Description: To determine the effect of ACZ885 versus placebo on other parameters of pulmonary function testing in patients with sarcoidosis at 24 weeks compared to baseline. Forced Expiratory Volume (FEV) in 1, 3, 6 seconds, predicted and forced expiratory flow 25-75%. Results expressed in change from baseline
Time Frame: Baseline, week 24
Population: Pharmacodynamic Analysis Set, with measure
Measure: Median (90% Confidence Interval); unit: Liter/second
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
Liter/second
  FEV in 1 Second: number analyzed (Participants) | 17 | 16
  FEV in 1 Second | -0.06 [-0.12 to 0.01] | 0.05 [-0.202 to 0.12]
  FEV in 3 seconds: number analyzed (Participants) | 17 | 16
  FEV in 3 seconds | -0.08 [-0.15 to 0.01] | 0.04 [-0.04 to 0.11]
  FEV in 6 seconds: number analyzed (Participants) | 17 | 16
  FEV in 6 seconds | -0.08 [-0.15 to 0.01] | 0.04 [-0.03 to 0.11]
  Predicted FEV: number analyzed (Participants) | 17 | 16
  Predicted FEV | -1.20 [-2.87 to 0.48] | 0.89 [-0.87 to 2.66]
  Forced Expiratory Flow 25-75%: number analyzed (Participants) | 17 | 16
  Forced Expiratory Flow 25-75% | -0.0 [-1.0 to 0.8] | 0.1 [-0.1 to 0.6]

6. Secondary Outcome: Change From Baseline in High Resolution Computed Tomography (HRCT) Scoring
Description: To determine the effect of ACZ885 versus placebo on HRCT of patients with sarcoidosis at 24 weeks compared to initial HRCT scan as measured by side-by-side comparison by blinded reviewers and HRCT scoring. HRCT score : sum of total parameters scores, each measured in different lung zones (right upper lobe; left upper lobe; right middle lobe; right lower lobe; left lower lobe). The extent of the disease is assessed for each zone to the nearest 10% of parenchymal surface: 0 (no disease) to 10 (91-100% disease).
Time Frame: Baseline, Week 24
Population: Pharmacodynamic Analysis Set, with measure
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale
  Parameter (unit): Mean of Consolidation: number analyzed (Participants) | 18 | 15
  Parameter (unit): Mean of Consolidation | 0.11 (0.21) | 0.00 (0.24)
  Parameter (unit): Mean of Fibrosis: number analyzed (Participants) | 18 | 15
  Parameter (unit): Mean of Fibrosis | 0.14 (0.20) | -0.26 (0.22)
  Parameter (unit): Mean of Ground Glass Opacities: number analyzed (Participants) | 18 | 15
  Parameter (unit): Mean of Ground Glass Opacities | 0.12 (0.39) | -0.21 (0.43)
  Parameter (unit): Mean of Linear Opacities: number analyzed (Participants) | 18 | 15
  Parameter (unit): Mean of Linear Opacities | -0.08 (0.04) | -0.00 (0.05)
  Parameter (unit): Mean of Nodule: number analyzed (Participants) | 18 | 15
  Parameter (unit): Mean of Nodule | 0.55 (0.57) | -0.46 (0.63)
  Parameter (unit): Mean of Total Sarcoidosis Score: number analyzed (Participants) | 18 | 15
  Parameter (unit): Mean of Total Sarcoidosis Score | 0.47 (1.04) | -0.79 (1.14)

7. Secondary Outcome: Change From Baseline Distance Walked as Assessed by the 6-minute Walk Test
Description: To determine the effect of ACZ885 versus placebo on the 6-minute walk test distance of patients with sarcoidosis at 12 and 24 weeks compared to baseline
Time Frame: Baseline, Week 12, and Week 24
Population: Pharmacodynamic Analysis Set, with measure
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
meter
  Baseline: number analyzed (Participants) | 4 | 4
  Baseline | 453.65 (98.643) | 502.36 (79.368)
  Week 12: number analyzed (Participants) | 4 | 4
  Week 12 | 471.57 (85.623) | 510.39 (99.555)
  Week 24: number analyzed (Participants) | 3 | 3
  Week 24 | 479.40 (95.212) | 511.74 (104.359)

8. Secondary Outcome: Change From Baseline of Additional [F-18]FDG-PET Outcomes
Description: To determine the effect of ACZ885 on additional [F-18]FDG-PET outcomes after 12 weeks of treatment compared to placebo. SUVmean: Mean standard uptake value for activity in the focal region volume SUVpeak: Mean standardized uptake value of a sphere (a diamater of approximately 1.2cm - to produce a 1-cm3-volume spherical Region of Interest (ROI) that has the highest average SUV with the lesion volume
Time Frame: Baseline, Week 12
Population: Pharmacodynamic Analysis Set, with measure
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change In SUVmean
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
Percentage of Change In SUVmean
  SUV mean lymph nodes: number analyzed (Participants) | 17 | 16
  SUV mean lymph nodes | -12.1 (8.09) | -4.77 (8.35)
  SUV mean lung parenchyma: number analyzed (Participants) | 16 | 15
  SUV mean lung parenchyma | -6.39 (9.00) | -3.87 (9.30)
  SUV mean extra thoracic region: number analyzed (Participants) | 4 | 7
  SUV mean extra thoracic region | -9.75 (15.23) | -15.2 (11.39)

9. Secondary Outcome: Change From Baseline in Other Parameters of Pulmonary Function Testing : Diffusion Capacity of Lung for CO
Description: To determine the effect of ACZ885 versus placebo on other parameters of pulmonary function testing in patients with sarcoidosis at 24 weeks compared to baseline.
Time Frame: Baseline, week 24
Population: Pharmacodynamic Analysis Set, with measure
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
mL/min/mmHg | -0.85 (1.740) | -1.05 (1.978)

10. Secondary Outcome: Change From Baseline in Other Parameters of Pulmonary Function Testing : Percent Predicted DLco, FEV1/FVC, FEV3/FVC, Percent Predicted Forced Expiratory Flow (FEF) 25-75, RV/TLC (Residual Volume /Total Lung Capacity)
Description: To determine the effect of ACZ885 versus placebo on other parameters of pulmonary function testing in patients with sarcoidosis at 24 weeks compared to baseline. Percent Predicted DLco (Diffusion Capacity of Lung for CO), FEV1/FVC, FEV3/FVC (forced expiratory volume in 1 or 3 seconds /forced vital capacity), percent Predicted FEF25-75, RV/TLC
Time Frame: Baseline, week 24
Population: Pharmacodynamic Analysis Set, with measure
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 20
percentage
  % Predicted DLco: number analyzed (Participants) | 13 | 14
  % Predicted DLco | -2.68 (5.082) | -2.71 (5.028)
  % FEV1/FVC: number analyzed (Participants) | 17 | 16
  % FEV1/FVC | 0.19 (3.549) | 0.73 (2.221)
  % FEV3/FVC: number analyzed (Participants) | 17 | 16
  % FEV3/FVC | -0.05 (2.617) | 0.21 (1.612)
  %Predicted FEF25-75: number analyzed (Participants) | 17 | 16
  %Predicted FEF25-75 | -0.94 (11.375) | 3.22 (5.485)
  % RV/TLC (Residual Volume /Total Lung Capacity): number analyzed (Participants) | 9 | 11
  % RV/TLC (Residual Volume /Total Lung Capacity) | 0.63 (3.106) | 0.23 (3.243)

ADVERSE EVENTS:
Time Frame: 40 months
Description: AE additional description
Groups:
- ACZ885 300 mg: ACZ885 300 mg
Arm/Group | ACZ885 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20 | 4/20
Other Adverse Events (participants affected / at risk) | 15/20 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 300 mg (N=20) | Placebo (N=20)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Atypical mycobacterium test positive (Investigations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 300 mg (N=20) | Placebo (N=20)
Ear pain (Ear and labyrinth disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 6 | 5
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 6
Pulpitis dental (Infections and infestations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT02888080/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT02888080/SAP_000.pdf